CLINICAL TRIAL: NCT07369453
Title: The Effects of Aerobic Exercise on Sleep Quality, Quality of Life, and Functional Status in Stroke Patients Treated With Botulinum Toxin for Upper Extremity Spasticity
Brief Title: Exercise to Improve Sleep and Quality of Life in Stroke Patients Receiving Botulinum Toxin Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bursa Yuksek Ihtisas Training and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Merve Yeni, Doctor, Department of Physical Medicine and Rehabilitation, Bursa Yuksek Ihtisas Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2011-KAEK-25 2021/08-12
Record Dates: First submitted 2025-12-23; First posted 2026-01-27 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Hemiplegia and/or Hemiparesis Following Stroke
Keywords: Botox; Aerobic Exercise; Spasticity; Sleep
MeSH Terms: conditions — Muscle Spasticity

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise Group (Experimental): Participants in this group received a supervised low- to moderate-intensity aerobic exercise program in addition to standard care. The aerobic exercise program was performed three times per week for four weeks, with 30-minute sessions consisting of warm-up, exercise, and cool-down periods. All participants also received botulinum toxin type A injections and conventional rehabilitation as part of routine clinical care.
  Interventions: Other: Aerobic exercise training using a cycle ergometer
- Control Group (No Intervention): Participants in this group received standard care only, consisting of botulinum toxin type A injections for upper extremity spasticity and conventional rehabilitation.

INTERVENTIONS:
Other: Aerobic exercise training using a cycle ergometer — A stationary cycling ergometer was used to deliver the supervised aerobic exercise intervention. The device was used for low- to moderate-intensity aerobic training at 40-60% of maximum heart rate, three sessions per week for four weeks, under medical supervision. The cycle ergometer is used solely as an exercise modality and is not the investigational product of the study.
  Arms: Aerobic Exercise Group

SUMMARY:
This study aimed to investigate the contribution of aerobic exercise programmes to improving sleep quality, quality of life, and functional status, alongside conventional rehabilitation, in stroke patients who had received botulinum toxin treatment for upper extremity spasticity.

DETAILED DESCRIPTION:
This randomized controlled trial included 62 chronic stroke patients receiving BTX-A injections for upper extremity spasticity. Participants were randomized into two groups: one that participated in a 4-week aerobic exercise program and a control group that received conventional rehabilitation without aerobic exercise. The primary outcomes were functional independence, upper extremity motor development, walking speed, sleep quality and quality of life.

ELIGIBILITY:
Inclusion Criteria:

* 62 patients aged 18-75 years who were planned for botulinum toxin treatment due to upper extremity spasticity following a stroke

Exclusion Criteria:

* Stroke patients who had BTX-A injections for lower extremity spasticity or had a Modified Ashworth Scale (MASH) score ≥ 2 for lower extremity spasticity,
* Uncontrolled diabetes, hypertension, cardiovascular diseases,
* Cognitive dysfunction,
* Flaccid stroke,
* Upper extremity disorders (fractures, frozen shoulder, arthritis, surgery),
* Pre-existing sleep disorders (obstructive sleep apnea, insomnia, parasomnia, narcolepsy, restless leg syndrome, or psychiatric disorders),
* Cancer diagnosis,
* Those who had received antispastic or antiepileptic treatment with dose changes in the last month

Ages: 18 Weeks to 75 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 56 (Actual)
Dates: Start 2021-09-15 (Actual); Primary Completion 2024-01-15 (Actual); Study Completion 2024-01-15 (Actual)

PRIMARY OUTCOMES:
Functional Recovery, Sleep, and Quality of Life Outcomes | From baseline to 12 weeks after starting the exercise program
  Health-related quality of life will be assessed using the Euroqol Quality of Life Scale, which evaluates mobility, selfcare, usual activities, pain and depression, with higher index values indicating better quality of life. Daytime sleepiness will be assessed using the Epworth Sleepiness Scale (0-24), where higher scores indicate greater sleepiness. Sleep quality will be evaluated using the Pittsburgh Sleep Quality Index (0-21), with higher scores indicating poorer sleep quality. Activities of daily living will be assessed using the Barthel Index (0-20). Functional independence will be evaluated using the Functional Independence Measure (18-126), with higher scores indicating greater independence. Neurological and motor recovery will be assessed using Brunnstrom stages, upper extremity motor function using the Fugl-Meyer Assessment of the Upper Extremity (0-66) and spasticity using the Modified Ashworth Scale. Functional exercise capacity will be assessed using the 6-Minute Walk Test.
Effects of Aerobic Exercise on Sleep Quality, Quality of Life, and Functional Status in Stroke Patients Treated with BTX-A for Upper Extremity Spasticity | From baseline to 12 weeks after starting the exercise program

CONTACTS AND LOCATIONS:
Locations (1):
- Bursa Yuksek Ihtisas Training and Research Hospital, Bursa, Turkey, Turkey (Türkiye)